CLINICAL TRIAL: NCT01043731
Title: Laparoscopic Transvaginal Hybrid Anterior Resection: a Prospective Data Collection
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Andreas Zerz, MD, Kantonal Hospital St. Gallen, Department of Visceral Surgery
Other Study IDs: EKSG09/151/2B
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-07

CONDITIONS: Sigmoid Diverticulitis (Hinchey I and II); Sigmoid Diverticulosis With Two or More Attacks of Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ginven indication for laparoscopic anterior resection
  Interventions: Procedure: Laparoscopic transvaginal hybrid anterior resection

INTERVENTIONS:
Procedure: Laparoscopic transvaginal hybrid anterior resection — Transvaginal Hybrid Anterior Resection: three 5mm trocars are placed transabdominally (one trans-umbilical, the other two in the lower abdomen). Identification of the inferior mesenteric vein and artery. Clipping of the vein. Then placement of a 12mm trocar through the posterior fornix of the vagina for stapling of the inferior mesenteric artery. After mobilisation of the colon descendens and the splenic flexure stapling of the proximal rectum through the 12mm trocar placed vaginally. Afterwards the colpotomy is performed and the mobilised left hemi-colon is extracted transvaginally. The proximal colonic resection is performed extracorporeally in the conventional fashion with placement of a purse-string suture and insertion of the circular stapling anvil into the proximal end of the bowel. The bowel is then replaced into the abdominal cavity. The colpotomy is then closed. A circular stapler is inserted transanally and the end-to-end anastomosis is performed.

SUMMARY:
Transvaginal hybrid procedures are of interest as an available NOTES-Procedure for the clinical routine. Few authors have demonstrated the feasibility and safety of such procedures (e.g. cholecystectomy) in selected patient collectives. In 2008 Lacy at al. published the experience with a transvaginal sigmoidectomy as a first in human report. The aim of this prospective data collection is to evaluate the feasibility and safety of the transvaginal hybrid anterior resection in the clinical routine.

Therefore all patients giving the informed consent to the transvaginal hybrid anterior resection will be included and assessed concerning feasibility to perform the transvaginal approach and complete the operation transvaginally.

ELIGIBILITY:
Inclusion Criteria:

* given informed consent
* sigmoid diverticulosis (two or more attacks)
* sigmoid diverticulitis (Hinchey I and II)

Exclusion Criteria:

* ASA IV
* emergency surgery
* liver-malfunction or coagulation disorders
* acute diverticulitis (Hinchey III and IV)
* malignancy
* acute vaginal infection
* refusal of mandatory preoperative gynecological examination
* pregnancy
* endometriosis
* previous surgery of colon and rectum
* strongly retroflexed uterus
* acute pelvic disorders, infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Given indication for laparoscopic anterior resection
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of the transvaginal operation | 30 days

SECONDARY OUTCOMES:
Long-term life quality and sexual dysfunction | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zerz, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of surgery, Sankt Gallen, Switzerland